CLINICAL TRIAL: NCT07044531
Title: DEVELOPMENT OF A NOVEL PEER RECOVERY SUPPORTER TRAINING PLATFORM TO DISSEMINATE EVIDENCE-BASED TRAINING AT SCALE
Brief Title: DEVELOPMENT OF A NOVEL PEER RECOVERY SUPPORTER TRAINING PLATFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thrive Digital Health, LLC (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4R44AA030953 (NIH); 4R44AA030953 (NIH)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Substance Use Disorders; Alcohol Use Disorders; Recovery Support Services; Peer Recovery Coaching
Keywords: Peer Recovery Support Services; Peer Recovery Coaching; Alcohol Use Disorders; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training as Usual (Active Comparator): Participants receive the standard, state-approved Connecticut Community on Addiction Recovery PRSS training program. No digital content or enhancements are provided.
  Interventions: Behavioral: Training-as-Usual (TAU)
- TDPP-A (Asynchronous Only) (Experimental): Participants access the Thrive Digital Peer Platform (TDPP) in fully asynchronous format. Content is self-paced, structured into 11 "Journeys" using the Connect → Grow → Apply model, and includes interactive modules and peer-led stories. No live facilitation is included.
  Interventions: Behavioral: TDPP-A (Asynchronous Platform)
- TDPP-Z (Asynchronous + Zoom) (Experimental): Participants use the TDPP asynchronous platform and also attend three live, facilitator-led group Zoom sessions designed to enhance skill development, application, and peer interaction. This hybrid model integrates digital learning with synchronous coaching.
  Interventions: Behavioral: TDPP-Z (Asynchronous + Zoom)

INTERVENTIONS:
Behavioral: Training-as-Usual (TAU) — Participants receive the standard Peer Recovery Supporter (PRS) training currently offered by CCAR. This training follows existing certification requirements and does not include any digital modules or facilitated teleconferencing components.
  Arms: Training as Usual
Behavioral: TDPP-A (Asynchronous Platform) — Participants engage with the Thrive Digital Peer Platform (TDPP), a fully asynchronous, self-paced online training program. The content includes 11 interactive modules structured using the Connect → Grow → Apply (CGA) learning framework, featuring peer stories, behavioral exercises, and scenario-based assessments.
  Arms: TDPP-A (Asynchronous Only)
Behavioral: TDPP-Z (Asynchronous + Zoom) — Participants use the same asynchronous TDPP platform as the TDPP-A group, with the addition of three live, facilitator-led Zoom sessions. These synchronous group sessions provide opportunities for applied learning, discussion, and skill reinforcement.
  Arms: TDPP-Z (Asynchronous + Zoom)

SUMMARY:
The focus of this study is to assess the effect on Peer Recovery Support Service providers of the fully asynchronous training platform (TDPP) and the TDPP with live zoom sessions on skill and adherence compared with training-as-usual.

DETAILED DESCRIPTION:
Thrive Digital Health ("TDH") is developing a novel Peer Recovery Support Services ("PRSS") training platform (the "TDPP") to standardize and scale the training of Peer Recovery Supporters. TDH was founded by the principals of two successful existing companies at the forefront of advancing PRSS, and benefits from the expertise of its CEO, who in addition to serving on the board of the Peer Recovery Center of Excellence, is a nationally recognized thought leader on PRSS training and implementation. The overarching goal of this Fasttrack project is to develop and test an evidence-based platform that will extend standards-based and empirically-supported Peer Recovery Support Services training and implementation across the country. Success in this endeavor will expand access to support services for recovery from alcohol and other substance use disorders, and help to address critical care gaps stemming from the treatment provider shortage currently impacting the nation. We hypothesize that this scalable platform, used by PRSS Trainers and Trainees, will be acceptable, feasible and usable, and will deliver a positive effect in terms of knowledge gain, adherence and skill in Phase I. In Phase II of this Fasttrack effort, we hypothesize that this platform will deliver superior training results among PRSS trainees in terms of adherence and skill versus training-as-usual. Our priority commercial goal is to bring this solution to market with organizations around the country seeking to build PRSS capacity, and we will accomplish this through the following Phase II specific aims: (1) Assess the effect on PRSS providers of the fully asynchronous TDPP and the TDPP with live zoom sessions on skill and adherence compared with training-as-usual; (2) Assess the effect of adding three live, interactive group teleconferencing sessions to the TDPP asynchronous content; (3) Conduct a pre-post study with a pilot population of PRSS provider trainees from another state to assess fidelity of implementation when content is localized for another state. The expected impact of this project is to substantially enhance TDH's ability to deliver effective PRSS training at scale, expanding access to recovery support services across the country. This capability holds promise to reduce negative health impacts at both an individual and societal level while reducing the total cost of providing treatment services.

ELIGIBILITY:
Inclusion Criteria: Eligible participants will be prospective PRSS providers residing in the U.S., ages 18 and over, with at least one year of continuous sobriety.

-

Exclusion Criteria: We will exclude individuals with eligibility questionnaire responses indicating: (a) an inability to read or speak English; (b) active suicidal ideation (PHQ-9, Item 9); (c) severe anxiety (GAD-7 >15); (d) significant medical illnesses, and; (e) unable to complete the baseline assessment or unavailable for computer and telephone follow-ups over the approximately ten month study period.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
YACS II Skill Adherence Score | Post-intervention (within 2 weeks of training completion)
  Assessed using the adapted Yale Adherence and Competence Scale II (YACS II), which measures skill adherence during simulated peer recovery support interactions. Each participant is scored by blinded, trained raters using a standardized coding protocol.

SECONDARY OUTCOMES:
System Usability Scale (SUS) Score | Immediately post-training
  Self-reported usability score using the System Usability Scale (SUS), a validated 10-item instrument that assesses the ease of use, satisfaction, and user experience of the TDPP platform.
Knowledge Gain (Knowledge Test) | Change from baseline to immediately post-training
  Improvement in participant scores on a knowledge test derived from the PRSS curriculum, administered pre- and post-training.
Intention to Use (UTAUT-2 scale) | Immediately post-training
  Assessed using the UTAUT-2 "Intention to Use" construct, scored on a 5-point Likert scale. Measures perceived likelihood of future platform use in practice.

OTHER OUTCOMES:
Self-Reported Satisfaction | Immediately post-training
  Participant-reported satisfaction with the training experience, assessed via a Likert-scale item ("How satisfied were you with the training experience overall?"). Scores range from 1 (not satisfied) to 5 (very satisfied).
Qualitative Feedback (Open-Ended Exit Interview) | Immediately post-training
  Participant reflections on their training experience, collected through a structured exit interview or open-text response field. Thematic content analysis will be used to identify emergent themes related to learning impact, perceived professionalism, and platform usability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pesce, JD/MBA, Principal Investigator — Thrive Digital Health, LLC
Locations (1):
- Thrive Digital Health, Solon, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided